CLINICAL TRIAL: NCT01291407
Title: A Phase I Study of S-1 in Combination With Radiotherapy in Locally Advanced or Recurrent Gastric Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Wang Xin, Dr., Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-012
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Gastrointestinal Neoplasms; Gastric Cancer
Keywords: Combined Modality; Gastric Cancer; Radiation Therapy; S-1
MeSH Terms: conditions — Gastrointestinal Neoplasms; Stomach Neoplasms | interventions — S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- S-1,peroral BID,capsule (Experimental)
  Interventions: Drug: S-1

INTERVENTIONS:
Drug: S-1 — S-1,30mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner.
  Other Names: an oral fluorinated pyrimidine combination
Drug: S-1 — S-1,40mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner.
  Other Names: an oral fluorinated pyrimidine combination
Drug: S-1 — S-1,50mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner
  Other Names: an oral fluorinated pyrimidine combination
Drug: S-1 — S-1,60mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner.
  Other Names: an oral fluorinated pyrimidine combination
Drug: S-1 — S-1,70mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner.
  Other Names: an oral fluorinated pyrimidine combination
Drug: S-1 — S-1,80mg/m2/d,peroral BID,in treatment days concurrently with radiation therapy in a standard manner.
  Other Names: an oral fluorinated pyrimidine combination

SUMMARY:
The purpose of this study is to determine maximum tolerated dose (MTD), dose limiting toxicities (DLT) and recommend a proper dose for our phase II study of S-1 when combined with radiation therapy for locally advanced or recurrent gastric cancer.

DETAILED DESCRIPTION:
This is a Phase I trial of S-1 given in treatment days with an oral dose from 30mg/m2/d to 80mg/m2/d, concurrently with radiation in patients with locally advanced or locally recurrent gastric cancer. Patients will be treated with external beam radiation therapy in a standard manner. S-1 will be administered for 6 dose levels,30/40/50/60/70/80mg/m2/d. Patients will be assessed for acute toxicities according to Common Toxicity Criteria for Adverse Effects (CTCAE)3.0.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven locally advanced gastric adenocarcinoma in patients undergoing R0, R1, R2 resection, or with unresectable or locoregional recurrent disease
* Any prior chemotherapy is allowed in this protocol.
* No distant metastasis in liver,lung,,bone,central nervous system(CNS),no peritoneal transplantation
* No prior abdominal or pelvic radiotherapy.
* Karnofsky performance status(KPS)≥ 70,predictive life span no less than 6 months
* Patients must have normal organ and marrow function as defined below:

  * Leukocytes greater than or equal to 3,000 G/L
  * Platelets: greater than or equal to 100,000/mm3
  * Hemoglobin:greater than or equal to 10g/L
  * Total bilirubin: within normal institutional limits
  * AST/ALT: less than or equal to 1.5 times the upper limit
  * Creatinine within normal upper limits
  * Informed consent
* Without any serious complications,such as hypertension,coronary artery disease,psychiatric history.

Exclusion Criteria:

* Patients with other cancer history except cervical carcinoma in situ and non-malignant melanoma skin cancer
* With any distant metastasis in liver,lung,,bone,CNS,or peritoneal transplantation
* History of allergic reactions attributed to similar chemical or biologic complex to S-1
* Uncontrolled illness including, but not limited to, active infection, symptomatic heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness
* History of myocardial infarction within the past 6 months or history of ventricular arrhythmia
* History of prior radiation to the abdomen
* Pregnant or lactating females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-11; Primary Completion 2013-08 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To define dose limited toxicities(DLT) of S-1, peroral BID, in treatment days concurrently with radiation therapy (RT) in locally advanced or recurrent gastric cancer. | up to 9 weeks
  Dose limited toxicities defined as below: leucopenia ≥4 neutropenia ≥ 4, anemia ≥ 3, thrombocytopenia ≥ 3, alanine aminotransferase/aspartate aminotransferase (AST) ≥ 3, alkaline phosphatase (ALT) ≥ 3, total bilirubin ≥ 3,blood urea nitrogen (BUN)/Cr ≥ 2,non-granular cell decreased fever ≥ 2, nausea/vomiting ≥ 2, fatigue ≥ 3, weight loss ≥ 3, diarrhea ≥ 3, abdominal pain ≥ 3, dysphagia ≥ 3, hand-foot syndrome ≥ 2, neurotoxicity ≥ 2.

SECONDARY OUTCOMES:
To define maximum tolerated dose(MTD) of S-1, peroral BID, in treatment days concurrently with radiation therapy | up to 9 weeks
  If 1 of 3 patients treated within a S-1 dose level experiences DLTs, 3 more patients will be treated at the same level. If a second patient experiences DLTs, then escalation will be stopped and the MTD is defined as the level below DLT dose level.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Jin, MD,PhD, Principal Investigator — Department of Radiation Oncology,Cancer Hospital and Institute,CAMS; Yexiong Li, MD,PhD, Principal Investigator — Department of Radiation Oncology,Cancer Hospital and Institute, CAMS
Locations (1):
- Department of Radiation Oncology, Cancer Hospital, Chinese Academy of Medical Sciences (CAMS) and Peking Union Medical College (PUMC), Beijing, China

REFERENCES:
- [Background] Parkin DM, Pisani P, Ferlay J. Global cancer statistics. CA Cancer J Clin. 1999 Jan-Feb;49(1):33-64, 1. doi: 10.3322/canjclin.49.1.33. PMID 10200776
- [Background] Taguchi T, Inuyama Y, Kanamaru R, Hasegawa K, Akazawa S, Niitani H, Furue H, Kurihara M, Ota K, Suga S, Ariyoshi Y, Takai S, Shimoyama T, Toge T, Takashima S, Sugimachi K, Hara Y, Fujita H, Kimura K, Saito T, Tsukagoshi S, Nakao I. [Phase I study of S-1. S-1 Study Group]. Gan To Kagaku Ryoho. 1997 Dec;24(15):2253-64. Japanese. PMID 9422070
- [Background] van Groeningen CJ, Peters GJ, Schornagel JH, Gall H, Noordhuis P, de Vries MJ, Turner SL, Swart MS, Pinedo HM, Hanauske AR, Giaccone G. Phase I clinical and pharmacokinetic study of oral S-1 in patients with advanced solid tumors. J Clin Oncol. 2000 Jul;18(14):2772-9. doi: 10.1200/JCO.2000.18.14.2772. PMID 10894878
- [Background] Cohen SJ, Leichman CG, Yeslow G, Beard M, Proefrock A, Roedig B, Damle B, Letrent SP, DeCillis AP, Meropol NJ. Phase I and pharmacokinetic study of once daily oral administration of S-1 in patients with advanced cancer. Clin Cancer Res. 2002 Jul;8(7):2116-22. PMID 12114411
- [Background] Chu QS, Hammond LA, Schwartz G, Ochoa L, Rha SY, Denis L, Molpus K, Roedig B, Letrent SP, Damle B, DeCillis AP, Rowinsky EK. Phase I and pharmacokinetic study of the oral fluoropyrimidine S-1 on a once-daily-for-28-day schedule in patients with advanced malignancies. Clin Cancer Res. 2004 Aug 1;10(15):4913-21. doi: 10.1158/1078-0432.CCR-04-0469. PMID 15297391
- [Background] Takahashi I, Kakeji Y, Emi Y, Sakurai M, Yonemura Y, Kimura Y, Maehara Y. S-1 in the treatment of advanced and recurrent gastric cancer: current state and future prospects. Gastric Cancer. 2003;6 Suppl 1:28-33. doi: 10.1007/s10120-003-0228-5. PMID 12775017
- [Background] Sakata Y, Ohtsu A, Horikoshi N, Sugimachi K, Mitachi Y, Taguchi T. Late phase II study of novel oral fluoropyrimidine anticancer drug S-1 (1 M tegafur-0.4 M gimestat-1 M otastat potassium) in advanced gastric cancer patients. Eur J Cancer. 1998 Oct;34(11):1715-20. doi: 10.1016/s0959-8049(98)00211-1. PMID 9893658
- [Background] Sugimachi K, Maehara Y, Horikoshi N, Shimada Y, Sakata Y, Mitachi Y, Taguchi T. An early phase II study of oral S-1, a newly developed 5-fluorouracil derivative for advanced and recurrent gastrointestinal cancers. The S-1 Gastrointestinal Cancer Study Group. Oncology. 1999 Oct;57(3):202-10. doi: 10.1159/000012032. PMID 10545788
- [Background] Koizumi W, Kurihara M, Nakano S, Hasegawa K. Phase II study of S-1, a novel oral derivative of 5-fluorouracil, in advanced gastric cancer. For the S-1 Cooperative Gastric Cancer Study Group. Oncology. 2000 Apr;58(3):191-7. doi: 10.1159/000012099. PMID 10765119
- [Background] Sakuramoto S, Sasako M, Yamaguchi T, Kinoshita T, Fujii M, Nashimoto A, Furukawa H, Nakajima T, Ohashi Y, Imamura H, Higashino M, Yamamura Y, Kurita A, Arai K; ACTS-GC Group. Adjuvant chemotherapy for gastric cancer with S-1, an oral fluoropyrimidine. N Engl J Med. 2007 Nov 1;357(18):1810-20. doi: 10.1056/NEJMoa072252. PMID 17978289
- [Background] Fujitani K, Tsujinaka T, Yamasaki H, Hirao M, Yoshida K, Kurokawa Y. Feasibility study of S-1 plus weekly docetaxel combined with concurrent radiotherapy in advanced gastric cancer refractory to first-line chemotherapy. Anticancer Res. 2009 Aug;29(8):3385-91. PMID 19661361
- [Background] Saikawa Y, Kubota T, Kumagai K, Nakamura R, Kumai K, Shigematsu N, Kubo A, Kitajima M, Kitagawa Y. Phase II study of chemoradiotherapy with S-1 and low-dose cisplatin for inoperable advanced gastric cancer. Int J Radiat Oncol Biol Phys. 2008 May 1;71(1):173-9. doi: 10.1016/j.ijrobp.2007.09.010. Epub 2007 Nov 8. PMID 17996385
- [Derived] Li N, Xiang X, Zhao D, Wang X, Tang Y, Chi Y, Yang L, Jiang L, Jiang J, Shi J, Liu W, Fang H, Tang Y, Chen B, Lu N, Jing H, Qi S, Wang S, Liu Y, Song Y, Li Y, Zhang L, Jin J. Preoperative versus postoperative chemo-radiotherapy for locally advanced gastric cancer: a multicenter propensity score-matched analysis. BMC Cancer. 2022 Feb 26;22(1):212. doi: 10.1186/s12885-022-09297-7. PMID 35219300